CLINICAL TRIAL: NCT04424641
Title: First-in-human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety of GEN1044 in Subjects With Malignant Solid Tumors
Brief Title: A Study on the Safety of GEN1044 (DuoBody®-CD3x5T4) in Patients With Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to MTD was reached
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1044-01; 2019-003998-26 (EudraCT Number); MOH_2020-07-26_008713 (Registry Identifier: Clinical Research Site - mytrial)
Record Dates: First submitted 2020-05-14; First posted 2020-06-11 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumor(s); Prostate Cancer; Esophageal Cancer; Triple Negative Breast Cancer (TNBC); Squamous Cell Carcinoma of Head and Neck (SCCHN); Non-small Cell Lung Cancer (NSCLC); Bladder Cancer; Uterine Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Esophageal Neoplasms; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Uterine Neoplasms | interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1044 (Experimental)
  Interventions: Biological: GEN1044 is an immunoglobulin G1 (IgG1) bispecific antibody targeting CD3 and 5T4.

INTERVENTIONS:
Biological: GEN1044 is an immunoglobulin G1 (IgG1) bispecific antibody targeting CD3 and 5T4. — GEN1044 will be administered intravenously in cycles of 21 days.
  Other Names: DuoBody®-CD3x5T4

SUMMARY:
The purpose of the trial is to evaluate the safety, determine the recommended Phase 2 dose (RP2D), and assess preliminary clinical activity of GEN1044 in patients with solid tumors.

DETAILED DESCRIPTION:
The trial is an open-label, multi-center safety trial of GEN1044. The trial consists of two parts: a dose-escalation part (Phase 1) and an expansion part (Phase 2a). The expansion part of the trial will be initiated once the RP2D has been determined from Phase 1.

ELIGIBILITY:
Key Inclusion Criteria:

Dose-escalation part:

• Patient with locally advanced or metastatic solid tumor(s) (excluding patients with primary central nervous system [CNS] tumors), who has experienced disease progression while on standard therapy or is intolerant of, or not eligible for, standard therapy.

Expansion part:

• Must have an advanced or metastatic, pathologically confirmed diagnosis of one of the following tumors: Uterine Cancer, Prostate Cancer, Esophageal Cancer, TNBC, SCCHN, NSCLC (both adenocarcinoma [ACC] and squamous cell carcinoma [SCC], Bladder Cancer.

Both parts:

* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for the trial, and is willing to participate in the trial prior to any trial related assessments or procedures.
* Must have measurable disease according to response assessment criteria relevant to the tumor type.
* Must have an Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-1 at Screening and on C1D1.
* A woman of reproductive potential must agree to use adequate contraception during the trial and for 4 months after the last GEN1044 administration. Adequate contraception is defined as highly effective methods of contraception.

Key Exclusion Criteria (both parts):

1. Has an uncontrolled intercurrent illness, including but not limited to:

   1. Ongoing or active infection requiring intravenous treatment with anti-infective therapy
   2. Symptomatic congestive heart failure (grade III or IV as classified by the New York Heart Association), unstable angina pectoris or cardiac arrhythmia.
   3. Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg, despite optimal medical management.
   4. Ongoing or recent evidence of significant autoimmune disease. Patients with a history of grade 3 or higher immune-related adverse events that led to treatment discontinuation.
   5. Patients with a prior history of myositis, Guillain-Barré syndrome, or myasthenia gravis of any grade.
   6. History of chronic liver disease or evidence of hepatic cirrhosis.
   7. History of non-infectious pneumonitis that has required steroids, or currently has pneumonitis.
   8. History of organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of GEN1044.
   9. Serious, non-healing wound, skin ulcer (of any grade), or bone fracture.
2. Any history of intracerebral arteriovenous malformation, cerebral aneurysm, new or symptomatic brain metastases or stroke.
3. Prior therapy:

   Radiotherapy: Radiotherapy within 14 days prior to first GEN1044 administration. Palliative radiotherapy will be allowed.
4. Treatment with an anti-cancer agent (within 28 days or after at least 5 half-lives of the drug, whichever is shorter), prior to GEN1044 administration. Toxicities from previous anti-cancer therapies that have not resolved.
5. Has a history of ≥ grade 2 cytokine release syndrome (CRS) with other CD3-based bispecifics, or a history of ≥ grade 3 allergic reactions to monoclonal antibody therapy as well as known or has known allergies, hypersensitivity, or intolerance to GEN1044 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Oliveri, MD, Study Director — Genmab
Locations (6):
- United States (2):
  - Tennesse Oncology, PLLC - Nashville, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Rigshospitalet (Copenhagen University Hospital), Copenhagen, Denmark
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid

REFERENCES:
- [Background] Kemper K, Gielen E, Boross P, Houtkamp M, Plantinga TS, de Poot SA, Burm SM, Janmaat ML, Koopman LA, van den Brink EN, Rademaker R, Verzijl D, Engelberts PJ, Satijn D, Sasser AK, Breij EC. Mechanistic and pharmacodynamic studies of DuoBody-CD3x5T4 in preclinical tumor models. Life Sci Alliance. 2022 Sep 8;5(11):e202201481. doi: 10.26508/lsa.202201481. Print 2022 Nov. PMID 36271507

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 48 participants signed the informed consent form of whom 37 received study drug. The Safety Committee decided to stop enrollment during the dose-escalation part and therefore the expansion part of trial never started. Consequently, results are available for only the dose-escalation part.
Groups:
- GEN1044 Doses 0.3/3/3 mg: Participants with locally advanced or metastatic non-central nervous system (CNS) solid tumor(s) received an IV infusion of GEN1044 weekly (0.3 mg on Cycle [C] 1 Day (D] 1 and 3 mg on C1D8 and C1D15) for the first 4 cycles (each cycle was 21 days), followed by every 3 weeks (Q3W) until the end of treatment.
- GEN1044 Doses 1/3/10 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 3 mg on C1D8, and 10 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- GEN1044 Doses 1/3/30 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 3 mg on C1D8, and 30 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- GEN1044 Doses 1/5/30 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 5 mg on C1D8, and 30 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- GEN1044 Doses 1/10/30 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 10 mg on C1D8, and 30 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- GEN1044 Doses 1/5/37.5 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 5 mg on C1D8, and 37.5 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- GEN1044 Doses 1/5/45 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 5 mg on C1D8, and 45 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- GEN1044 Doses 1/3/60 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (1 mg on C1D1, 3 mg on C1D8, and 60 mg on C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
Period: Overall Study
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
Started | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6
Not completed — Death | 1 | 2 | 3 | 0 | 3 | 0 | 1 | 2
Not completed — Sponsor decision | 0 | 2 | 3 | 7 | 2 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of study drug. Participants were classified according to the assigned dose level cohort.
Groups:
- GEN1044 Doses 0.3/3/3 mg: Participants with locally advanced or metastatic non-CNS solid tumor(s) received an IV infusion of GEN1044 weekly (0.3 mg on C1D1 and 3 mg on C1D8 and C1D15) for the first 4 cycles (each cycle was 21 days), followed by Q3W until the end of treatment.
- Total: Total of all reporting groups
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg | Total
Number analyzed (Participants) | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.0 (NA) — Standard deviation was not derived as only one participant was evaluated for this arm. | 61.3 (12.89) | 60.4 (11.21) | 59.3 (8.18) | 62.3 (5.79) | 52.0 (8.49) | 55.8 (15.71) | 54.2 (15.29) | 58.4 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 3 | 4 | 1 | 2 | 3 | 19
  Male | 0 | 2 | 4 | 4 | 2 | 1 | 2 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 2 | 5 | 1 | 0 | 0 | 2 | 11
  Unknown or Not Reported | 0 | 4 | 5 | 2 | 5 | 2 | 4 | 4 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 4 | 6 | 5 | 6 | 2 | 4 | 5 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: The DLT was defined as Grade (G) >= 3 cytokine release syndrome or immune effector cell-associated neurotoxicity syndrome; any G3 or 4 hematologic and non-hematologic toxicity (with exceptions defined by the protocol); laboratory abnormality that required clinically significant medical intervention, led to hospitalization, persisted for >1 week, or resulted in a drug-induced liver injury; G3 or 4 febrile neutropenia; liver toxicity defined by Hy's law; any treatment-related toxicity that caused treatment discontinuation during Cycle 1; or any G5 toxicity.
Time Frame: From Day 1 to Day 21 of first cycle
Population: Dose-determining set (DDS) included all participants who received at least 1 dose of study drug during the dose-escalation part, and who met the minimum exposure criterion and had sufficient safety evaluations or experienced a DLT during the first 21 days of dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
Number analyzed (Participants) | 1 | 4 | 4 | 3 | 2 | 0 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 1 |  | 3 | 3

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) is defined as an AE that meets one of the following criteria: fatal or life-threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; medically significant (an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above [medical and scientific judgment must be exercised in deciding whether an AE is 'medically significant']); required inpatient hospitalization or prolongation of existing hospitalization. A TEAE is defined as an AE occurring or worsening between the first dose of GEN1044 and 30 days after the last dose received.
Time Frame: Day 1 through Day 263 (corresponding to maximum observed duration)
Population: Safety set included all participants who received at least 1 dose of study drug. Participants were classified according to the assigned dose level cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
Number analyzed (Participants) | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6
Participants
  Any TEAE | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6
  Any TESAE | 1 | 1 | 3 | 5 | 4 | 1 | 3 | 5

3. Primary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Number of participants with laboratory values of Grade >= 3 by NCI-CTCAE v5.0 are reported. The NCI-CTCAE is a descriptive terminology that is used for gradings (Grade 1-5) of Adverse Events (AEs) and of laboratory values; the latter being summarized here.
  This table reports laboratory values graded only on the numerical value of the reported parameter and is therefore not graded by symptoms or signs. The abnormal laboratory values assessed by the investigator as being AEs are reported also in the AE table.
  In case a participant reported multiple severity grades for a laboratory value, only the maximum grade was used.
Time Frame: Day 1 through Day 263 (corresponding to maximum observed duration)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
Number analyzed (Participants) | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6
Participants
  Lymphocyte count decreased | 1 | 4 | 7 | 4 | 5 | 2 | 2 | 6
  Lipase increased | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2
  Serum amylase increased | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1
  Hypomagnesemia | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  Creatinine increased | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Anemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Hypokalemia | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hypoalbuminemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gamma-glutamyl transferase increased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR)
Description: The radiological evaluation based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) was performed by investigator using computed tomography (CT) scan/ magnetic resonance imaging (MRI) scan/ positron emission tomography (PET) scan. The CR was defined as disappearance of all target and non-target lesions and all pathological lymph nodes must have decreased to < 10 mm in short axis. The PR was defined as at least a 30% decrease in the sum of the longest diameters of target lesions taking as reference the baseline sum of longest diameters.
Time Frame: Day 1 through Day 233
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
Number analyzed (Participants) | 1 | 4 | 7 | 7 | 6 | 2 | 4 | 6
Participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs) Positive to GEN1044
Description: The detection and titer characterization of ADAs was performed using validated, specific, and sensitive electrochemiluminescence immunoassay (ECLIA) methods. Number of participants with ADA positive post baseline to GEN1044 are reported.
Time Frame: Day 1 through Day 263 (predose on Day 1 of Cycles 1, 2, 3, 5, 7, and then on Day 1 of every 4 cycles thereafter, end of treatment [EOT], and 30 days after last study drug)
Population: Immunogenicity analysis set included all participants who received at least 1 dose of study drug and had evaluable immunogenicity samples.
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
Number analyzed (Participants) | 1 | 4 | 7 | 3 | 6 | 2 | 4 | 4
Participants | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: For AEs: Day 1 through Day 263 (corresponding to maximum observed duration); For All-cause mortality: From date of inform consent form through Day 263 (corresponding to maximum observed duration)
Description: The adverse events were evaluated per the safety set. The safety set included all participants who received at least 1 dose of GEN1044. Participants were classified according to the assigned dose level cohort. One (1) death in the 1/10/30 mg reporting group was recorded 5 days after the patient withdrew trial consent.
Arm/Group | GEN1044 Doses 0.3/3/3 mg | GEN1044 Doses 1/3/10 mg | GEN1044 Doses 1/3/30 mg | GEN1044 Doses 1/5/30 mg | GEN1044 Doses 1/10/30 mg | GEN1044 Doses 1/5/37.5 mg | GEN1044 Doses 1/5/45 mg | GEN1044 Doses 1/3/60 mg
All-Cause Mortality (participants affected / at risk) | 1/1 | 2/4 | 3/7 | 0/7 | 4/6 | 0/2 | 1/4 | 2/6
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/4 | 3/7 | 5/7 | 4/6 | 1/2 | 3/4 | 5/6
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 7/7 | 7/7 | 6/6 | 2/2 | 4/4 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEN1044 Doses 0.3/3/3 mg (N=1) | GEN1044 Doses 1/3/10 mg (N=4) | GEN1044 Doses 1/3/30 mg (N=7) | GEN1044 Doses 1/5/30 mg (N=7) | GEN1044 Doses 1/10/30 mg (N=6) | GEN1044 Doses 1/5/37.5 mg (N=2) | GEN1044 Doses 1/5/45 mg (N=4) | GEN1044 Doses 1/3/60 mg (N=6)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 1 (6) | 0 (0) | 1 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 2 (10) | 3 (13) | 3 (9) | 0 (0) | 2 (9) | 3 (9)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (5)
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEN1044 Doses 0.3/3/3 mg (N=1) | GEN1044 Doses 1/3/10 mg (N=4) | GEN1044 Doses 1/3/30 mg (N=7) | GEN1044 Doses 1/5/30 mg (N=7) | GEN1044 Doses 1/10/30 mg (N=6) | GEN1044 Doses 1/5/37.5 mg (N=2) | GEN1044 Doses 1/5/45 mg (N=4) | GEN1044 Doses 1/3/60 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (7) | 6 (23) | 4 (15) | 5 (13) | 1 (2) | 4 (15) | 4 (12)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 5 (9) | 4 (6) | 4 (6) | 1 (1) | 3 (6) | 5 (10)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (8) | 5 (10) | 2 (4) | 5 (11) | 0 (0) | 4 (8) | 4 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (2) | 0 (0) | 1 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (5) | 2 (2) | 3 (3) | 1 (2) | 2 (3) | 2 (3)
Fatigue (General disorders) | 0 (0) | 4 (7) | 4 (8) | 0 (0) | 4 (7) | 1 (1) | 2 (3) | 1 (2)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (4) | 3 (10) | 2 (6) | 3 (4) | 3 (14) | 2 (4) | 2 (4) | 4 (14)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive Protein Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (5) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (5)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 2 (5)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hot Flush (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Upon review and evaluation of the overall safety profile and safety signals of GEN1044 during the dose-escalation part, the Safety Committee decided to stop further enrollment and the Sponsor decided to stop the compound development. Hence, the expansion part of the trial was never initiated, and while a majority of the pharmacokinetic (PK) samples from the dose-escalation part were quantified, the PK parameters were not calculated due to termination of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 12 months but less than 18 months from the end of study (database lock). The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04424641/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT04424641/SAP_001.pdf